CLINICAL TRIAL: NCT01198301
Title: Gene Expression Profiling of Metastatic Breast Cancer Predict the Therapeutic Response to Chemotherapy
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Ren, Director, Peking University Cancer Hospital & Institute
Other Study IDs: GEP
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: Metastatic Breast Neoplasms; Gene Expression Profiling; Drug Therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the tissue will be obtained by core niddle biopsy.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators want to develop a gene expression profile the for prediction the chemotherapeutic response of patients with metastatic breast cancer.

DETAILED DESCRIPTION:
1. Metastatic breast cancer tissue is obtained from core needle biopsies pretreatment and is flash frozen and stored at -70℃ until processing.
2. After patients received docetaxel combination thiotepa for two cycles, response is assessed using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines. Degree of response is used to divide the cancers into two groups-sensitive and resistant tumours.
3. The gene expression in metastatic breast cancer tissue sample is detected by microarray to screen gene markers that are differently expressed between groups
4. Statistical analysis is performed using unsupervised hierarchical cluster.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be histologically confirmed with metastatic breast cancer;
* Patients who had completed the planned chemotherapy regimen with no major protocol violation;
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* At least one measurable lesion;
* Normal cardiac, hepatic, renal and bone marrow functions;
* Life expectancy ≥3 months;
* Discontinuity of previous chemotherapy for a minimum of 4 weeks.

Exclusion Criteria:

* previous history of other malignancies;
* previous surgery history on the needle biopsy organ;
* Central nervous system metastases;
* Serious or uncontrolled concurrent medical illness.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with metastatic breast cancer treated by Docetaxel-based chemotherapy
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Chemotherapy response | four-months
  Response to chemotherapy is assessed using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines

SECONDARY OUTCOMES:
Time to disease progression | six months
  Time to disease progression is measured from the date therapy is initiated to the date of documented disease progression.
Overall survival | one year
  Overall survival is measured from the date therapy is initiated to the date of death or final follow-up.
clinical benefit response | six months to one year
  clinical benefit response include CR,PR,SD

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; Jun Ren, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China